CLINICAL TRIAL: NCT05375383
Title: Assessment of Colonisation of Probiotic Bacterium Streptococcus Salivarius in the Oral Cavity
Brief Title: Microbial Colonization of Oral Probiotics
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: BLIS Technologies Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: BLTCT2022/3
Record Dates: First submitted 2022-05-11; First posted 2022-05-16 (Actual); Last update posted 2022-05-16 (Actual); Status verified 2022-05

CONDITIONS: Microbial Colonization
Keywords: Streptococcus salivarius K12; Probiotic; microbial colonization; oral probiotic; lozenges; powder; prebiotic; Streptococcus salivarius M18
MeSH Terms: conditions — Communicable Diseases

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of the 12 groups consuming powder or lozenges containing Streptococcus salivarius K12 or S. salivarius M18 with or without prebiotic:
  Probiotic S. salivarius K12 lozenges Probiotic S. salivarius K12 lozenges containing prebiotic A Probiotic S. salivarius K12 lozenges containing prebiotic B Probiotic S. salivarius K12 lozenges containing prebiotic A and B
  Probiotic S. salivarius K12 powder Probiotic S. salivarius K12 powder containing prebiotic A Probiotic S. salivarius K12 powder containing prebiotic B Probiotic S. salivarius K12 powder containing prebiotic A and B
  Probiotic S. salivarius M18 lozenges Probiotic S. salivarius M18 lozenges containing prebiotic A Probiotic S. salivarius M18 lozenges der containing prebiotic B Probiotic S. salivarius M18 + lozenges containing prebiotic A and B
Who Masked: Participant, Investigator
Masking Description: A staff member not part of the study group will be assigned to distribute blinded samples. The participant or the investigators will not be aware of the dose groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (12):
- Streptococcus salivarius K12 lozenge (Active Comparator): Streptococcus salivarius K12 lozenge
  Interventions: Dietary Supplement: Streptococcus salivarius K12 lozenge
- Probiotic S. salivarius K12 lozenges containing prebiotic A (Active Comparator): Streptococcus salivarius K12 lozenge with prebiotic
  Interventions: Dietary Supplement: Probiotic S. salivarius K12 lozenges containing prebiotic A
- Probiotic S. salivarius K12 lozenges containing prebiotic B (Active Comparator): Streptococcus salivarius K12 lozenge with prebiotic
  Interventions: Dietary Supplement: Probiotic S. salivarius K12 lozenges containing prebiotic B
- Probiotic S. salivarius K12 lozenges containing prebiotic A and B (Active Comparator): Streptococcus salivarius K12
  Interventions: Dietary Supplement: Probiotic S. salivarius K12 lozenges containing prebiotics A and B
- Probiotic S. salivarius K12 powder (Active Comparator): Streptococcus salivarius K12 powder
  Interventions: Dietary Supplement: Probiotic S. salivarius K12 powder
- Probiotic S. salivarius K12 powder containing prebiotic A (Active Comparator): Streptococcus salivarius K12 powder with prebiotic
  Interventions: Dietary Supplement: Probiotic S. salivarius K12 powder containing prebiotic A
- Probiotic S. salivarius K12 powder containing prebiotic B (Active Comparator): Streptococcus salivarius K12 powder with prebiotic
  Interventions: Dietary Supplement: Probiotic S. salivarius K12 powder containing prebiotic B
- Probiotic S. salivarius K12 powder containing prebiotic A and B (Active Comparator): Streptococcus salivarius K12 powder with prebiotic
  Interventions: Dietary Supplement: Probiotic S. salivarius K12 powder containing prebiotics A and B
- Probiotic S. salivarius M18 lozenges (Active Comparator): Streptococcus salivarius M18 lozenge
  Interventions: Dietary Supplement: Probiotic S. salivarius M18 lozenges
- Probiotic S. salivarius M18 lozenges containing prebiotic A (Active Comparator): Streptococcus salivarius M18 lozenge with prebiotic
  Interventions: Dietary Supplement: Probiotic S. salivarius M18 lozenges containing prebiotic A
- Probiotic S. salivarius M18 lozenges der containing prebiotic B (Active Comparator): Streptococcus salivarius M18 lozenge with prebiotic
  Interventions: Dietary Supplement: Probiotic S. salivarius M18 lozenges containing prebiotic B
- Probiotic S. salivarius M18 + lozenges containing prebiotic A and B (Active Comparator): Streptococcus salivarius M18 lozenge with prebiotic
  Interventions: Dietary Supplement: Probiotic S. salivarius M18 + lozenges containing prebiotic A and B

INTERVENTIONS:
Dietary Supplement: Streptococcus salivarius K12 lozenge — In this study, a lozenge will be evaluated for its potential of delivering probiotic Streptococcus salivarius K12 to the oral cavity.
  Arms: Streptococcus salivarius K12 lozenge
Dietary Supplement: Probiotic S. salivarius K12 lozenges containing prebiotic A — In this study, a lozenge containing a prebiotic will be evaluated for its potential of delivering probiotic Streptococcus salivarius K12 to the oral cavity.
  Arms: Probiotic S. salivarius K12 lozenges containing prebiotic A
Dietary Supplement: Probiotic S. salivarius K12 lozenges containing prebiotic B — In this study, a lozenge containing a prebiotic will be evaluated for its potential of delivering probiotic Streptococcus salivarius K12 to the oral cavity.
  Arms: Probiotic S. salivarius K12 lozenges containing prebiotic B
Dietary Supplement: Probiotic S. salivarius K12 lozenges containing prebiotics A and B — In this study, a lozenge containing two prebiotics will be evaluated for its potential of delivering probiotic Streptococcus salivarius K12 to the oral cavity.
  Arms: Probiotic S. salivarius K12 lozenges containing prebiotic A and B
Dietary Supplement: Probiotic S. salivarius K12 powder — In this study, a powder will be evaluated for its potential of delivering probiotic Streptococcus salivarius K12 to the oral cavity
  Arms: Probiotic S. salivarius K12 powder
Dietary Supplement: Probiotic S. salivarius K12 powder containing prebiotic A — In this study, a powder containing a prebiotic will be evaluated for its potential of delivering probiotic Streptococcus salivarius K12 to the oral cavity
  Arms: Probiotic S. salivarius K12 powder containing prebiotic A
Dietary Supplement: Probiotic S. salivarius K12 powder containing prebiotic B — In this study, a powder containing a prebiotic will be evaluated for its potential of delivering probiotic Streptococcus salivarius K12 to the oral cavity
  Arms: Probiotic S. salivarius K12 powder containing prebiotic B
Dietary Supplement: Probiotic S. salivarius K12 powder containing prebiotics A and B — In this study, a powder containing two prebiotics will be evaluated for its potential of delivering probiotic Streptococcus salivarius K12 to the oral cavity
  Arms: Probiotic S. salivarius K12 powder containing prebiotic A and B
Dietary Supplement: Probiotic S. salivarius M18 lozenges — In this study, a lozenge containing will be evaluated for its potential of delivering probiotic Streptococcus salivarius M18 to the oral cavity.
  Arms: Probiotic S. salivarius M18 lozenges
Dietary Supplement: Probiotic S. salivarius M18 lozenges containing prebiotic A — In this study, a lozenge containing a prebiotic will be evaluated for its potential of delivering probiotic Streptococcus salivarius M18 to the oral cavity.
  Arms: Probiotic S. salivarius M18 lozenges containing prebiotic A
Dietary Supplement: Probiotic S. salivarius M18 lozenges containing prebiotic B — In this study, a lozenge containing a prebiotic will be evaluated for its potential of delivering probiotic Streptococcus salivarius M18 to the oral cavity.
  Arms: Probiotic S. salivarius M18 lozenges der containing prebiotic B
Dietary Supplement: Probiotic S. salivarius M18 + lozenges containing prebiotic A and B — In this study, a lozenge containing two prebiotics will be evaluated for its potential of delivering probiotic Streptococcus salivarius M18 to the oral cavity.
  Arms: Probiotic S. salivarius M18 + lozenges containing prebiotic A and B

SUMMARY:
The aim of this study is to evaluate the colonization efficacy of probiotic lozenges and powders containing specific prebiotics in healthy adults

DETAILED DESCRIPTION:
This is a double-blind, randomized controlled colonization pilot study with no cross over to evaluate the colonization efficacy of lozenges and powders containing two different commercially available probiotic bacteria (S. salivarius K12 ) or S. salivarius M18 with or without 2 different prebiotic sugars or their combinations.

Participants will be randomly assigned to one of the 12 groups consuming probiotic lozenge or powder containing Streptococcus salivarius K12 or S. salivarius M18 with or without prebiotics (e.g. sugars that may promote probiotic activity) over a seven day period. Saliva samples will be collected at predetermined time points pre and post intervention. Colonisation efficacy will be determined by enumerating the probiotic in the saliva samples using standard microbiological techniques.

ELIGIBILITY:
Inclusion criteria:

1. Male or Female 18y - 80y age
2. In general good health 18 - 80 years of age.
3. Practice good oral hygiene.

Exclusion criteria:

1. Have a history of autoimmune disease or are immunocompromised.
2. Are on concurrent antibiotic therapy or regular antibiotic use within last 1 week
3. History of allergy (e.g. dairy).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-06-15 (Estimated); Primary Completion 2022-08-31 (Estimated); Study Completion 2022-09-15 (Estimated)

PRIMARY OUTCOMES:
Change in microbial colonization from baseline (Day 0) to 1 hour for S. salivarius K12 lozenges | 1 hour
  Study will determine the change in microbial colonization efficacy of Streptococcus salivarius K12 with or without prebiotics from a lozenge format. The statistical analysis (e.g. Students t-test) will be carried out to compare the participants data from baseline to one hour after later across different formulations with the level of significance of p≤0.05.Overall colonization based on percentage of population colonized for different interventions will also be analyzed average and standard deviation functions using appropriate statistical analysis software (e.g. Microsoft Excel).
Change in microbial colonization from baseline (Day 0) to 8 hours or S. salivarius K12 lozenges | 8 hour
  Study will determine the change in microbial colonization efficacy of Streptococcus salivarius K12 with or without prebiotics from a lozenge format. The statistical analysis (e.g. Students t-test) will be carried out to compare the participants data from baseline to eight hours after later across different formulations with the level of significance of p≤0.05.Overall colonization based on percentage of population colonized for different interventions will also be analyzed average and standard deviation functions using appropriate statistical analysis software (e.g. Microsoft Excel).
Change in microbial colonization from baseline (Day 0) to 24 hours or S. salivarius K12 lozenges | 24 hour
  Study will determine the change in microbial colonization efficacy of Streptococcus salivarius K12 with or without prebiotics from a lozenge format. The statistical analysis (e.g. Students t-test) will be carried out to compare the participants data from baseline to 24 hours after later across different formulations with the level of significance of p≤0.05.Overall colonization based on percentage of population colonized for different interventions will also be analyzed average and standard deviation functions using appropriate statistical analysis software (e.g. Microsoft Excel).
Change in microbial colonization from baseline (Day 0) to 48 hours or S. salivarius K12 lozenges | 48 hour
  Study will determine the change in microbial colonization efficacy of Streptococcus salivarius K12 with or without prebiotics from a lozenge format. The statistical analysis (e.g. Students t-test) will be carried out to compare the participants data from baseline to 48hours after later across different formulations with the level of significance of p≤0.05.Overall colonization based on percentage of population colonized for different interventions will also be analyzed average and standard deviation functions using appropriate statistical analysis software (e.g. Microsoft Excel).
in microbial colonization from baseline (Day 0) to 1 hour for S. salivarius K12 powder format | 1 hour
  Study will determine the change in microbial colonization efficacy of Streptococcus salivarius K12 with or without prebiotics from a powder format. The statistical analysis (e.g. Students t-test) will be carried out to compare the participants data from baseline to one hour after later across two different formulations with the level of significance of p≤0.05.Overall colonization based on percentage of population colonized for different interventions will also be analyzed average and standard deviation functions using appropriate statistical analysis software (e.g. Microsoft Excel).
in microbial colonization from baseline (Day 0) to 8 hour for S. salivarius K12 powder format | 8 hours
  Study will determine the change in microbial colonization efficacy of Streptococcus salivarius K12 with or without prebiotics from a powder format. The statistical analysis (e.g. Students t-test) will be carried out to compare the participants data from baseline to 8 hours after later across two different formulations with the level of significance of p≤0.05.Overall colonization based on percentage of population colonized for different interventions will also be analyzed average and standard deviation functions using appropriate statistical analysis software (e.g. Microsoft Excel).
in microbial colonization from baseline (Day 0) to 24 hours for S. salivarius K12 powder format | 24 hours
  Study will determine the change in microbial colonization efficacy of Streptococcus salivarius K12 with or without prebiotics from a powder format. The statistical analysis (e.g. Students t-test) will be carried out to compare the participants data from baseline to 24 hours after later across two different formulations with the level of significance of p≤0.05.Overall colonization based on percentage of population colonized for different interventions will also be analyzed average and standard deviation functions using appropriate statistical analysis software (e.g. Microsoft Excel).
in microbial colonization from baseline (Day 0) to 48 hours for S. salivarius K12 powder format | 48 hours
  Study will determine the change in microbial colonization efficacy of Streptococcus salivarius K12 with or without prebiotics from a powder format. The statistical analysis (e.g. Students t-test) will be carried out to compare the participants data from baseline to 48 hours after later across two different formulations with the level of significance of p≤0.05.Overall colonization based on percentage of population colonized for different interventions will also be analyzed average and standard deviation functions using appropriate statistical analysis software (e.g. Microsoft Excel).
Change in microbial colonization from baseline (Day 0) to 1 hour for S. salivarius M18 lozenges | 1 hour
  Study will determine the change in microbial colonization efficacy of Streptococcus salivarius M18 with or without prebiotics from a lozenge format. The statistical analysis (e.g. Students t-test) will be carried out to compare the participants data from baseline to one hour after later across different formulations with the level of significance of p≤0.05.Overall colonization based on percentage of population colonized for different interventions will also be analyzed average and standard deviation functions using appropriate statistical analysis software (e.g. Microsoft Excel).
Change in microbial colonization from baseline (Day 0) to 8 hours for S. salivarius M18 lozenges | 8 hour
  Study will determine the change in microbial colonization efficacy of Streptococcus salivarius M18 with or without prebiotics from a lozenge format. The statistical analysis (e.g. Students t-test) will be carried out to compare the participants data from baseline to 8 hour after later across different formulations with the level of significance of p≤0.05.Overall colonization based on percentage of population colonized for different interventions will also be analyzed average and standard deviation functions using appropriate statistical analysis software (e.g. Microsoft Excel).
Change in microbial colonization from baseline (Day 0) to 24 hours for S. salivarius M18 lozenges | 24 hour
  Study will determine the change in microbial colonization efficacy of Streptococcus salivarius M18 with or without prebiotics from a lozenge format. The statistical analysis (e.g. Students t-test) will be carried out to compare the participants data from baseline to 24 hour after later across different formulations with the level of significance of p≤0.05.Overall colonization based on percentage of population colonized for different interventions will also be analyzed average and standard deviation functions using appropriate statistical analysis software (e.g. Microsoft Excel).
Change in microbial colonization from baseline (Day 0) to 48 hours for S. salivarius M18 lozenges | 48 hour
  Study will determine the change in microbial colonization efficacy of Streptococcus salivarius M18 with or without prebiotics from a lozenge format. The statistical analysis (e.g. Students t-test) will be carried out to compare the participants data from baseline to 48 hour after later across different formulations with the level of significance of p≤0.05.Overall colonization based on percentage of population colonized for different interventions will also be analyzed average and standard deviation functions using appropriate statistical analysis software (e.g. Microsoft Excel).

CONTACTS AND LOCATIONS:
Overall Officials: John D Hale, PhD, Study Director — Blis Technologies Ltd; Rohit Jain, PhD, Principal Investigator — Blis Technologies Ltd, Dunedin, New Zealand; John R Tagg, PhD, Principal Investigator — Blis Technologies Ltd, Dunedin, New Zealand
Locations (1):
- Blis Technologies Ltd, Dunedin, Otago, New Zealand

IPD SHARING:
Plan to Share IPD: Yes
Data and information included in the Protocol and Clinical Study Report will be shared to other researchers and/or in publications in due course.
Supporting Information: Study Protocol, CSR
Time Frame: Study report 3 months after the completion of the study.
Access Criteria: Summary study report will be shared by Principal investigator upon request if not published in public literature.

REFERENCES:
- [Background] Hyink O, Wescombe PA, Upton M, Ragland N, Burton JP, Tagg JR. Salivaricin A2 and the novel lantibiotic salivaricin B are encoded at adjacent loci on a 190-kilobase transmissible megaplasmid in the oral probiotic strain Streptococcus salivarius K12. Appl Environ Microbiol. 2007 Feb;73(4):1107-13. doi: 10.1128/AEM.02265-06. Epub 2006 Dec 28. PMID 17194838
- [Background] Burton JP, Chilcott CN, Wescombe PA, Tagg JR. Extended Safety Data for the Oral Cavity Probiotic Streptococcus salivarius K12. Probiotics Antimicrob Proteins. 2010 Oct;2(3):135-44. doi: 10.1007/s12602-010-9045-4. PMID 26781236
- [Background] Gregori G, Righi O, Risso P, Boiardi G, Demuru G, Ferzetti A, Galli A, Ghisoni M, Lenzini S, Marenghi C, Mura C, Sacchetti R, Suzzani L. Reduction of group A beta-hemolytic streptococcus pharyngo-tonsillar infections associated with use of the oral probiotic Streptococcus salivarius K12: a retrospective observational study. Ther Clin Risk Manag. 2016 Jan 19;12:87-92. doi: 10.2147/TCRM.S96134. eCollection 2016. PMID 26855579
- [Background] Di Pierro F, Adami T, Rapacioli G, Giardini N, Streitberger C. Clinical evaluation of the oral probiotic Streptococcus salivarius K12 in the prevention of recurrent pharyngitis and/or tonsillitis caused by Streptococcus pyogenes in adults. Expert Opin Biol Ther. 2013 Mar;13(3):339-43. doi: 10.1517/14712598.2013.758711. Epub 2013 Jan 4. PMID 23286823
- [Background] Di Pierro F, Colombo M, Zanvit A, Rottoli AS. Positive clinical outcomes derived from using Streptococcus salivarius K12 to prevent streptococcal pharyngotonsillitis in children: a pilot investigation. Drug Healthc Patient Saf. 2016 Nov 21;8:77-81. doi: 10.2147/DHPS.S117214. eCollection 2016. PMID 27920580
- [Background] Di Pierro F, Colombo M, Giuliani MG, Danza ML, Basile I, Bollani T, Conti AM, Zanvit A, Rottoli AS. Effect of administration of Streptococcus salivarius K12 on the occurrence of streptococcal pharyngo-tonsillitis, scarlet fever and acute otitis media in 3 years old children. Eur Rev Med Pharmacol Sci. 2016 Nov;20(21):4601-4606. PMID 27874935
- [Background] Di Pierro F, Zanvit A, Nobili P, Risso P, Fornaini C. Cariogram outcome after 90 days of oral treatment with Streptococcus salivarius M18 in children at high risk for dental caries: results of a randomized, controlled study. Clin Cosmet Investig Dent. 2015 Oct 3;7:107-13. doi: 10.2147/CCIDE.S93066. eCollection 2015. PMID 26491371
- [Background] Bardellini E, Amadori F, Gobbi E, Ferri A, Conti G, Majorana A. Does Streptococcus Salivarius Strain M18 Assumption Make Black Stains Disappear in Children? Oral Health Prev Dent. 2020 Apr 3;18(2):161-164. doi: 10.3290/j.ohpd.a43359. PMID 32099975